CLINICAL TRIAL: NCT03546491
Title: A Clinical Study to Evaluate Anti-Plaque Benefit of a Gel in a Modified- 4 Day Plaque Model
Brief Title: Evaluate Dental Plaque Benefit of a Preventive Treatment Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018009
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preventive Gel (Experimental): 0.4% stannous fluoride
  Interventions: Drug: Preventive Gel
- Marketed Control (Active Comparator): 0.243 % Sodium Fluoride
  Interventions: Drug: Marketed Control

INTERVENTIONS:
Drug: Preventive Gel — 0.4% Stannous Fluoride
  Arms: Preventive Gel
Drug: Marketed Control — 0.243% Sodium Fluoride
  Arms: Marketed Control

SUMMARY:
The objective of the study is to evaluate anti-plaque efficacy of a preventive treatment gel in a modified 4-day plaque model.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be 18 years of age or older;
* Agree not to participate in any other oral/dental product studies during the study;
* Agree to delay any elective dentistry (including dental prophylaxis) until the study has been completed;
* Agree to refrain from the use of any non-study oral hygiene products (subjects who are regular flossers will be allowed to floss during acclimation and wash-out periods);
* Agree to use an oral hygiene product that contains stannous fluoride;
* Agree to refrain from any form of non-specified oral hygiene during the treatment period, including the use of products such as floss, toothpicks for plaque removal, and chewing gum;
* Agree to refrain from any oral hygiene, eating and drinking after 11:00 PM the evening before plaque measurements on Day 0 and Day 4 of the treatment periods;
* Agree to return for all scheduled visits and follow study procedures;
* Possess a minimum of 20 natural teeth with scorable facial and lingual surfaces, of which at least 4 are molars; and,
* Be in good general health, as determined by the Investigator/designee based on a review of the health history/update for participation in the study.

Exclusion Criteria:• Have a medical condition requiring pre-medication prior to dental procedures;

* Have taken antibiotics within 2 weeks of the acclimation period or anticipate taking antibiotics at any time during the study;
* Have a history of allergies or hypersensitivity to dyes or dentifrices that contain stannous fluoride;
* Have removable or orthodontic appliances which interfere with obtaining 20 gradable teeth;
* Have previously demonstrated an inability to comply with study visit requirements;
* Have rampant caries, open or untreated caries, severe gingivitis or advanced periodontitis requiring prompt treatment; or,
* Present with any disease or condition(s) that could be expected to interfere with examination procedures or the subject's safe completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Health Science Center, Mason, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: This was a single center, controlled, examiner-blind, randomized, 2-treatment, 3-period cross-over 4-day partial brushing plaque study. Each participant received Test product 1 (0.4% stannous fluoride preventive gel), and Test product 2 (marketed 0.243% sodium fluoride toothpaste). All subjects saw each test product at least 1 time, for the third period, each subject saw either Test product 1 or Test product 2 for a second time.
Period: Overall Study
Arm/Group | Overall Study
Started | 32
Recieved Test Product 1 (This was a 2 treatment, 3 period crossover design, each subject saw one treatment twice.) | 32
Received Test Product 2 (This was a 2 treatment, 3 period crossover design, each subject saw one treatment twice.) | 32
Completed | 30
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This was a controlled, examiner-blind, randomized, 2-treatment, 3-period cross-over 4-day partial brushing plaque study.
Arm/Group | Overall Study
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Asian | 2
  Ethnicity: Black or African American | 5
  Ethnicity: Not Reported | 1
  Ethnicity: White Caucasian | 24
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Turesky Modified Quigley-Hein Index at Day 4
Description: The Turesky Modified Quigley-Hein Index was scored on six surfaces (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual and mesiolingual) to assess plaque on all gradable teeth. Whole mouth average plaque scores were calculated for each subject and tooth surfaces by totaling the scores and dividing by the number of gradable sites examined. the scoring criteria is below; (0) No Plaque; (1) Separate flecks of plaque at the cervical margin; (2) A thin, continuous band of plaque (up to 1 mm) at the cervical margin; (3) A band of plaque wider than 1 mm, but covering less than one third of the side of the crown of the tooth; (4) Plaque covering at least one third, but less than two thirds of the side of the crown of the tooth; (5) Plaque covering two thirds or more of the side of the crown of the tooth.
Time Frame: Day 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Gel | Marketed Control
Number analyzed (Participants) | 32 | 32
score on a scale | 1.83 (0.055) | 1.96 (0.055)

2. Secondary Outcome: Mean Turesky Modified Quigley-Hein Index at Baseline
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Preventive Gel | Marketed Control
Number analyzed (Participants) | 32 | 32
score on a scale | 2.19 (0.07) | 2.22 (0.07)

3. Secondary Outcome: Digital Plaque Imaging
Description: Total percent dental plaque area
Time Frame: Day 4
Measure: Mean (Standard Error); unit: percentage of plaque area
Groups:
- Preventive Gel: 0.4% stannous fluoride Preventive Gel
Arm/Group | Preventive Gel | Marketed Control
Number analyzed (Participants) | 32 | 32
percentage of plaque area | 8.14 (0.871) | 10.95 (0.871)

4. Secondary Outcome: Overall Baseline Mean Digital Plaque Imaging
Description: Total percent dental plaque area
Time Frame: Baseline
Measure: Mean (Standard Error); unit: percentage of plaque area
Groups:
- Marketed Control: 0.243% Sodium fluoride toothpaste
Arm/Group | Preventive Gel | Marketed Control
Number analyzed (Participants) | 32 | 32
percentage of plaque area | 6.57 (1.18) | 7.29 (1.18)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entire duration of the study for each intervention.
Arm/Group | Preventive Gel | Marketed Control
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 8/32 | 6/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preventive Gel (N=32) | Marketed Control (N=32)
Irritation Gum (Gastrointestinal disorders) | 2 | 2
Irritation Lip (Gastrointestinal disorders) | 0 | 1
Desquamation Oral (Gastrointestinal disorders) | 1 | 1
Irritation Mouth (Gastrointestinal disorders) | 5 | 2
Herpetic Lesion Oral (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03546491/Prot_SAP_000.pdf